CLINICAL TRIAL: NCT02996357
Title: Specific Factors Associated With the Development of Incontinence- Associated Dermatitis (IAD) in ICU Patients Suffering From Fecal Incontinence: Matched Case Control Study
Brief Title: Risk Factors for Incontinence-Associated Dermatitis (IAD) in ICU Patients Suffering From Fecal Incontinence
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016/0883
Record Dates: First submitted 2016-08-26; First posted 2016-12-19 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Irritant Contact Dermatitis; Diaper Rash; Incontinence-associated Dermatitis
Keywords: Incontinence-associated dermatitis; Risk factor; Intensive care unit; Prevention
MeSH Terms: conditions — Dermatitis, Irritant; Diaper Rash

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with IAD Category 2 (red skin with skin breakdown)
- Controls: Patients with IAD Cat. 0 (at risk, no redness and skin intact)

SUMMARY:
This study aims to identify patient characteristics associated with the development of Incontinence-Associated Dermatitis (IAD) category 2 (skin erosion due to incontinence).

380 ICU patients suffering of fecal incontinence will be included in the study. Data on 19 possible risk factors will be collected at one point in time by the research team. Different sources and methods will be used to collect patient data: skin assessment, patient record, direct patient observation, routine blood samples.

DETAILED DESCRIPTION:
Incontinence is a widespread problem in all health care settings. Prevalence figures of incontinence vary around 20.0% of all hospitalized patients. In acute and critical care units the proportion of patients with fecal incontinence may rise up to 33.0%.

One of the main complications of incontinence is inflammation of the skin in the genital and anal region, also known as incontinence-associated dermatitis (IAD). IAD is defined as skin inflammation manifested as redness with or without blistering, erosion, or loss of skin barrier function that occurs as a consequence of chronically or repeated exposure of the skin to urine or faeces.

A range of skin care products and procedures for the prevention of IAD exists. In order to provide cost-effective IAD prevention, it's important to target preventive skin care interventions to patients at risk of IAD.

The aims of this study are:

1. To identify specific factors associated with the development of Incontinence- Associated Dermatitis (IAD) in a recognized high risk patient population (ICU patients suffering from fecal incontinence)
2. To develop and statistically validate patient profiles being associated with high risk for IAD development

This study is a matched case control study. The cases are defined as patients with IAD Cat. 2 (red skin with skin breakdown). The controls are defined as patients with IAD Cat. 0 (at risk, no redness and skin intact). The patient will be matched for fecal incontinence.

In total, 380 ICU patients suffering from fecal incontinence will be included. 19 possible risk factors will be studied.

All data will be collected at one point in time by the research team. Different sources and methods will be used to collect patient data: skin assessment, patient record, direct patient observation, routine blood samples.

Specific IAD risk factors will be determined by applying univariate and multivariate binary logistic regression modeling.

ELIGIBILITY:
Inclusion Criteria:

* Being admitted to the intensive care unit
* Being fecal incontinent (=unintentional loss of stool)

Exclusion Criteria:

* Being < 18 years
* No contact possible between skin en stool at the perianal region (e.g. due to enteral stoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care unit, with fecal incontinence (a known risk for IAD Cat. 2 development) will be sampled. The presence of fecal incontinence (any type) will be used as the only variable for matching (as not to reduce the possibility to interfere with associated risk factors).
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation score (APACHE II) | 1 day
Presence of mechanical ventilation | Up to six days
Presence of dialysis | Up to six days
Presence of infection | Up to six days
  Leucocyten count and white blood cell count
Presence of fever | Up to six days
  temperature > 38.0°C
Presence of inadequate arterial oxygen pressure | Up to six days
  PaO2 < 80mmHg
Administration of antibiotics | Up to six days
Administration of steroids | Up to six days
Presence of malnutrition | Up to six days
  Measured by serum albumin level
Presence of diabetes | Up to six days
Use of continence products (diapers, underpads) | Up to six days
Use of washing without water (wipes, skin cleansers) | Up to six days
Presence of urinary incontinence | Up to six days
Presence of diarrhea | Up to six days
  Measured by Bristol Stool Chart
Presence of Clostridium difficile | Up to six days
Presence of mechanical chafing | Up to six days
Presence of low hemoglobin level | Up to six days
Presence of enteral nutrition | Up to six days
Presence of diminished cognitive awareness | Up to six days
  Measured by Glasgow Coma Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, PhD, Principal Investigator — University Ghent
Locations (19):
- Belgium (19):
  - Onze-Lieve-Vrouwziekenhuis Aalst, Aalst
  - ZiekenhuisNetwerk Antwerpen, Antwerp
  - AZ Monica, Deurne
  - Ziekenhuis Oost-Limburg, Genk
  - Algemeen Ziekenhuis Jan Palfijn, Ghent
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - Universitair Ziekenhuis Brussel, Jette
  - Algemeen Ziekenhuis Groeninge, Kortrijk
  - Universitaire Ziekenhuizen van de K.U. Leuven, Leuven
  - Algemeen Ziekenhuis Sint Maarten, Mechelen
  - Algemeen Ziekenhuis Delta, Roeselare
  - AZ Nikolaas, Sint-Niklaas
  - Algemeen Ziekenhuis Sint-Augustinus, Veurne
  - O.L.V. van Lourdesziekenhuis, Waregem
  - De Gasthuiszusters Antwerpen, Wilrijk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beeckman D, Van Damme N, Schoonhoven L, Van Lancker A, Kottner J, Beele H, Gray M, Woodward S, Fader M, Van den Bussche K, Van Hecke A, De Meyer D, Verhaeghe S. Interventions for preventing and treating incontinence-associated dermatitis in adults. Cochrane Database Syst Rev. 2016 Nov 10;11(11):CD011627. doi: 10.1002/14651858.CD011627.pub2. PMID 27841440
- [Background] Beeckman D, Van Lancker A, Van Hecke A, Verhaeghe S. A systematic review and meta-analysis of incontinence-associated dermatitis, incontinence, and moisture as risk factors for pressure ulcer development. Res Nurs Health. 2014 Jun;37(3):204-18. doi: 10.1002/nur.21593. Epub 2014 Apr 3. PMID 24700170
- See also: Website of the research group — http://www.ucvvgent.be